CLINICAL TRIAL: NCT05678881
Title: A Phase 1b Randomized, Double-Blind, Placebo Controlled, Crossover Study to Evaluate the Safety, Tolerability, and Efficacy of Two Doses of RLS103 (Inhaled Dry Powder Cannabidiol [CBD]) in a Clinical Model of Photosensitive Epilepsy
Brief Title: Safety, Tolerability, and Efficacy of RLS103 in a Clinical Model of Photosensitive Epilepsy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Receptor Life Sciences (Industry)
Collaborators: The Epilepsy Study Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RC2022-02
Record Dates: First submitted 2022-12-22; First posted 2023-01-10 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High dose RLS103 (Experimental): 8 mg CBD inhaled dry powder
  Interventions: Drug: High dose RLS103
- Placebo (Placebo Comparator): placebo inhaled dry powder
  Interventions: Drug: placebo inhaled powder
- Low dose RLS103 (Experimental): 4 mg CBD inhaled dry powder (open label)
  Interventions: Drug: Low dose RLS103

INTERVENTIONS:
Drug: High dose RLS103 — 8 mg CBD inhaled powder
  Arms: High dose RLS103
Drug: placebo inhaled powder — placebo inhaled powder
  Arms: Placebo
Drug: Low dose RLS103 — 4 mg CBD inhaled powder (open label)
  Arms: Low dose RLS103

SUMMARY:
The purpose of this study is to evaluate RLS103 for safety and suppression of the epileptic photoparoxysmal response compared to placebo.

DETAILED DESCRIPTION:
Approximately 5 subjects with a known stable photoparoxysmal response (PPR) on EEG, will be administered high dose RLS103 and placebo in a blinded, randomized, crossover design. Patient EEG responses will be compared between RLS103 and placebo. An additional low dose RLS103 may be administered to each patient in an open label period.

On study days, several procedures and intermittent photic stimulation (IPS) assessments will be performed at pre-determined times over the course of the day. After the subject completes both treatment visits, the blinded IPS data will be reviewed and analyzed by the Sponsor and the Epilepsy Study Consortium, Inc. If the blinded data on the 2 treatment days indicates a differential response, a decision will be made whether the subject will be asked to continue in the open label phase. The open label phase will consist of one visit, lasting 1 day.

ELIGIBILITY:
Inclusion Criteria:

* Must sign an informed consent form (ICF) indicating that they understand the purpose of the study and the procedures required for the study; and are willing to participate in the study and attend all visits and requirements.
* Individuals age 18-65 years, inclusive.
* A history of a photoparoxysmal response on EEG with or without a diagnosis of epilepsy for which subjects are on 0-3 concomitant antiseizure medications (ASMs).
* At least 3 of the EEGs performed during the Screening Visit must have a reproducible IPS-induced photoparoxysmal response (PPR) on EEG of ≥3 points on a frequency assessment scale in the same eye condition.
* Subjects in otherwise good health (with the exception of epilepsy), as determined by the PI via the medical history, a physical examination and screening laboratory investigations.
* A body mass index (BMI) between 17.5 to 42
* Participants agree to refrain from strenuous exercise the day before Screening and during the day prior to treatment days.
* Females of childbearing potential must commit to the consistent and correct use of an effective method of birth control throughout the study and must also have negative pregnancy test results at all visits prior to investigational product (IP) administration. Effective methods of contraception include surgical sterilization of the subject, condoms with spermicide, diaphragm with spermicide, hormonal contraceptive agents (oral, transdermal, or injectable), or implantable contraceptive devices.
* Negative viral serology test results for hepatitis B and C virus.
* Must have no medical contraindication to CBD, including known allergies or hypersensitivities to CBD or the excipients in RLS103.
* Must demonstrate the ability to use the inhaler correctly through a training tool (BluHale).
* Must have the ability and willingness to attend the necessary clinic visits.

Exclusion Criteria:

* A history of non-epileptic seizures (e.g. metabolic, structural or pseudo-seizures).
* Females who are pregnant or lactating.
* Individuals of reproductive potential who do not agree to use effective birth-control methods.
* Any clinically significant laboratory abnormality which, in the opinion of the investigator, will exclude the subject from the study.
* An active CNS infection, demyelinating disease, degenerative neurological disease or any CNS disease deemed to be progressive during the course of the study that may confound the interpretation of the study results.
* Any clinically significant psychiatric illness, psychological or behavioral problems which, in the opinion of the investigator, would interfere with the subject's ability to participate in the study.
* A history of alcoholism, drug abuse, or drug addiction within the past 12 months.
* Subjects who are suffering from clinically significant active liver disease, porphyria or with a family history of severe hepatic dysfunction indicated by abnormal liver function tests greater than 3 times the upper limit of normal (AST and ALT).
* Subjects who have participated in any other trials involving an investigational product or device within 30 days of screening or longer as required by local regulations.
* Subjects receiving more than 3 concomitant ASMs for their epilepsy.
* In the opinion of the Investigator, has a significant risk for suicidal behavior during the course of their participation in the study, or
* At Screening (Visit 1): the subject scores "yes" on items 1 or 2 in the Suicidal Ideation section of the Columbia-Suicide Severity Rating Scale (C-SSRS) with reference to a 6-month period prior to Screening; or
* At Screening (Visit 1): the subject has had 1 or more suicidal attempts with reference to a 2-year period prior to Screening; or
* At Visit 2 or Visit 3: the subject scores "yes" on items 1 or 2 in the Suicidal Ideation section of the C-SSRS with reference to Screening; or
* The subject is considered to be an imminent danger to themself or others.
* Currently using marijuana, marijuana cigarettes, cannabis-related products, THC (e.g. dronabinol, Marinol, Syndros) or CBD (e.g. Epidiolex or any over-the-counter CBD-containing product); or have used any of these products within 3 weeks prior to Screening (at the discretion of the Investigator in consultation with the Sponsor, to be confirmed by a urine drug test at Screening).
* Any history of pulmonary disease, including bronchospastic respiratory disease (bronchial asthma), or chronic obstructive pulmonary disease.
* Clinically significant abnormal values for spirometry, or hematology, serum chemistry, or urinalysis at Screening as deemed appropriate by the Investigator, including:
* Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >1.5 × the upper limit of normal (ULN)
* Total bilirubin >1.5 × ULN (isolated bilirubin >1.5 ×ULN is acceptable if total bilirubin and direct bilirubin <35%)
* Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Received an investigational medicinal product within 30 days or 5 half-lives prior to Baseline, whichever is longer.
* Fever (body temperature >38°C) or symptomatic viral or bacterial infection within 2 weeks prior to Screening, including confirmed active COVID-19.
* Had major surgery (general anesthetic) in the last 3 months or minor surgery (local anesthetic) in the last 1 month prior to Screening or have any pre-planned surgery or procedures that would interfere with the conduct of the study.
* Is an employee of the Investigator or study site, with direct involvement in the proposed study or other studies under the direction of that Investigator or study site, as well as family members of the employees or the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | 1 week (between Visits 2 and 3)
  Number and severity of treatment emergent serious adverse events (TESAEs), treatment emergent adverse events (TEAEs),and adverse events (AEs) leading to discontinuation from the study.
Change in PPR | 1 week (between Visits 2 and 3)
  Change in the PPR range in subjects receiving RLS103 compared to placebo

SECONDARY OUTCOMES:
Change in concomitant plasma ASM levels | 1 week (between Visits 2 and 3)
  Plasma concentrations of concomitant anti-seizure medications (ASMs) during administration of RLS103 as compared to the placebo days
CBD pharmacokinetics | 1 hour
  Plasma concentration of CBD at 2, 10, 30, and 60 minutes after inhalation

IPD SHARING:
Plan to Share IPD: No